CLINICAL TRIAL: NCT02278705
Title: Primary Care Clinical Practice Elements and Improving Overweight Children's Weight Status
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1K23HL118152-01A1 Aim 1; 1K23HL118152-01A1 (NIH)
Record Dates: First submitted 2014-10-24; First posted 2014-10-30 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Overweight; Childhood Obesity
Keywords: childhood obesity; childhood overweight; primary care; weight management
MeSH Terms: conditions — Overweight; Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Weight-status improved: Cases, termed, "weight-status improved," are defined as children whose BMI percent relative to their age/sex-specific BMI at the 95th percentile decreases from one visit to the next; and from one well-child visit to the next well-child (or primary-care visit approximately 9-18 months later).
  Interventions: Other: Attention to BMI; Other: Attention to high-BMI-related Medical Risk; Other: No attention to high BMI or high-BMI-related medical risk
- Weight-status unchanged/worse: Controls are defined as children whose BMI percent relative to their age/sex-specific BMI at the 95th percentile remains unchanged or increases from one visit to the next; and from one well-child visit to the next well-child (or primary-care visit approximately 9-18 months later).
  Interventions: Other: Attention to BMI; Other: Attention to high-BMI-related Medical Risk; Other: No attention to high BMI or high-BMI-related medical risk

INTERVENTIONS:
Other: Attention to BMI — Evidence (using electronic health record data) denoting provider attention to about high BMI.
  Other Names: BMI
Other: Attention to high-BMI-related Medical Risk — Evidence (using electronic health record data) denoting provider attention to high-BMI-related medical risk, including from high blood pressure/hypertension, cholesterol/dyslipidemia, blood sugar/diabetes, liver enzymes/fatty liver, and low vitamin D/vitamin-D deficiency.
  Other Names: Medical Risk
Other: No attention to high BMI or high-BMI-related medical risk — Lack of evidence (using electronic health record data) denoting provider attention to high BMI or high-BMI-related medical risk.
  Other Names: No BMI/Medical-Risk Attention

SUMMARY:
The purpose of this study is to identify whether specific clinical practices-including attention to body-mass-index (BMI) screening/overweight/obesity, medical risk (from conditions associated with overweight/obesity such as high blood pressure), and following up to reassess progress-will improve the weight status of overweight school-age children.

DETAILED DESCRIPTION:
The aim of this study is to identify specific clinical practice elements in pediatric primary care that predict improvement in weight status among overweight school-age children. Pediatricians are well-suited to regularly assess and treat school-age children who are overweight. Well-child visits present an important opportunity to assess and treat overweight children. Strategies are needed to maximize the effectiveness of this opportunity. Although the American Academy of Pediatrics endorses recommendations by the United States Preventive Services Task Force that clinicians screen for overweight, assess medical/behavior risk, and use a staged treatment approach that includes frequent reassessment, it is unclear whether these practices, when used in primary care, impact whether children make lifestyle changes or improve their weight status. It is essential to identify specific clinical practice elements and communication strategies associated with weight-status improvement in overweight children, to maximize the effectiveness of primary-care weight-management interventions. The investigators hypothesize that, during primary-care visits with overweight 6-12-year-old children, attention to high BMI, medical risk (from weight-related comorbidities such as high blood pressure), and reassessing progress (defined as having a primary-care visit with evidence of attention to BMI or completing a referral to a weight-management specialist or nutritionist) will be associated with improvement in weight status (assessed as decrease in percent overweight (percentage above the age/sex-specific 95th BMI percentile) at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 year-old children with ≥2 visits
* valid height and weight data at each visit
* BMI ≥85th percentile at the first visit

Exclusion Criteria:

* children <6 and >12 years old
* no valid height and weight data at two visits
* BMI <85th percentile at all 6-12 year-old well child visits

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Overweight 6-12 year-old children followed by pediatricians at community-based and academic primary-care clinics. A random sample of controls will be matched to cases by age, gender, race/ethnicity, BMI-percentile category, and clinic site.
Sampling Method: Probability Sample
Enrollment: 7192 (Actual)
Dates: Start 2009-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
weight-status improvement | From one visit to the next and from one well-child visit to the next
  Children with a decrease in BMI percent relative to the age/sex-specific BMI at the 95th percentile

CONTACTS AND LOCATIONS:
Overall Officials: Christy B Turer, MD, MHS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern and Children's Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Turer CB, Montano S, Lin H, Hoang K, Flores G. Pediatricians' communication about weight with overweight Latino children and their parents. Pediatrics. 2014 Nov;134(5):892-9. doi: 10.1542/peds.2014-1282. Epub 2014 Oct 13. PMID 25311599
- [Background] Turer CB, Mehta M, Durante R, Wazni F, Flores G. Parental perspectives regarding primary-care weight-management strategies for school-age children. Matern Child Nutr. 2016 Apr;12(2):326-38. doi: 10.1111/mcn.12131. Epub 2014 Apr 10. PMID 24720565
- [Background] Upperman C, Palmieri P, Lin H, Flores G, Turer CB. What do parents want for their children who are overweight when visiting the paediatrician? Obes Sci Pract. 2015 Oct;1(1):33-40. doi: 10.1002/osp4.5. Epub 2015 Sep 10. PMID 28580163
- [Background] Turer CB, Upperman C, Merchant Z, Montano S, Flores G. Primary-Care Weight-Management Strategies: Parental Priorities and Preferences. Acad Pediatr. 2016 Apr;16(3):260-6. doi: 10.1016/j.acap.2015.09.001. Epub 2015 Sep 26. PMID 26514648
- [Background] Turer CB, Barlow SE, Montano S, Flores G. Discrepancies in Communication Versus Documentation of Weight-Management Benchmarks: Analysis of Recorded Visits With Latino Children and Associated Health-Record Documentation. Glob Pediatr Health. 2017 Feb 6;4:2333794X16685190. doi: 10.1177/2333794X16685190. eCollection 2017. PMID 28239625